CLINICAL TRIAL: NCT05567588
Title: A Phase II,Single-arm Study to Evaluate the Safety and Efficacy of Pembrolizumab and Stereotactic Radiotherapy (SBRT) in Patients Advanced Metastatic Renal Clear Cell Carcinoma.
Brief Title: Pembrolizumab Plus Radiotherapy for Advanced Renal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2022-248
Record Dates: First submitted 2022-10-02; First posted 2022-10-05 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma
Keywords: pembrolizumab; stereotactic radiotherapy
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pembrolizumab + RT (5 fractions, 8 Gy) + Pembrolizumab (Experimental): Pembrolizumab will be started. Stereotactic Body Radiation Therapy will be given before the 2nd course of pembrolizumab and pembrolizumab will be continued.
  Pembrolizumab will continue until progression as per immune related response criteria (irRC).
  Interventions: Combination Product: Drug: Pembrolizumab

INTERVENTIONS:
Combination Product: Drug: Pembrolizumab — 200mg(body weight >75kg) or 100mg(body weight≤75kg) given intravenously over 30 minutes day 1 of every 3 week cycle until progression as per immune related response criteria.
  Other Names: Keytruda

SUMMARY:
This study is designed as a phase-II proof of clinical trial to investigate if a treatment strategy where stereotactic body radiation therapy (SBRT) is given with pembrolizumab is sufficiently active to warrant further investigation in randomized phase II or III studies. Metastatic renal cell cancer (mRCC) patients with PD-1 expressing immune cells are more likely to have larger more aggressive tumours and reduced survival. Pembrolizumab is designed to directly block the interaction between PD-1 and its ligands, PD-L1 and PD-L2. SBRT will be given to the 1-5 most clinically significant lesions after the 1nd course of pembrolizumab treatment in an effort to improve the activity of pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years at the time of signing informed consent;
* ECOG score of 0 or 1;
* Histologically confirmed, advanced ccRCC of stage IV (AJCC 8);
* Life expectancy of more than 12 weeks;
* Evidence of measurable metastatic kidney cancer according to RECIST 1.1 criteria. Patients should have an adequate number of non-irradiated metastatic sites in order to adequately assess the activity of the pembrolizumab therapy;
* If central nervous system (CNS) metastases are treated before inclusion and the patient's neurological system is present Return of symptoms to baseline levels (except for signs or symptoms associated with CNS therapy)At least 14 days, such patients may be included. In addition, patients must stop taking glucocorticoids or prednisone in a stable dose and ≤ 10 mg per day;
* Main organ function meets the following criteria within 7 days before treatment:

  1. blood examination criteria (in the state without blood transfusion within 14 days): ① Hemoglobin(HB) ≥ 70 g/L; ② Absolute Neutrophil Count(ANC) ≥ 1.0×109/L; ③ Platelet (PLT) ≥ 60×109/L.
  2. Biochemical examination shall meet the following criteria: ① total bilirubin within 1.5×the upper limit of normal(ULN); ② serum transaminase≤2.5×the Upper Limit of Normal(ULN), If associated with liver metastasis, serum transaminase≤5.0×the Upper Limit of Normal(ULN);③ serum creatine ≤ 1.5 x Upper Limit of Normal(ULN),creatinine clearance rate ≥ 60ml/min;
* Women of childbearing age should agree to use contraception (e. g. intrauterine device, contraceptive or condom) within 6 months after study completion, the pregnancy test results (serum or urine) within 7 days before enrolment must be negative;
* Men should agree that contraception must be used during and within 6 months of the end of the study period;
* With consent and have signed the informed consent, willing and able to comply with the planned visits, research treatment, laboratory tests, and other experimental procedures.

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2;
* Any active or recently diagnosed clear or suspected autoimmune disorder disease, or symptoms requiring glucocorticoids (> 10 mg/day) or immunosuppressive drugs for systemic therapy;
* Active brain metastases and/or cancerous meningitis;
* Has had a prior monoclonal antibody within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier;
* Has more than one previous chemotherapy,targeted small molecule therapy, or radiation therapy within 2 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent;
* Diagnosed with immunodeficiency within 2 weeks prior to study or being treated with systemic glucocorticoids or any other form of immunosuppressive therapy;
* Have a positive history of human immunodeficiency virus (HIV) test or have acquired immunodeficiency syndrome (AIDS);
* Has known active Hepatitis B or Hepatitis C;
* Has a known additional malignancy that is progressing or requires active treatment;
* Have interstitial lung disease, active pulmonary infectious pneumonia, or grade 3 or higher pneumonia;
* Patients with mental or physical illnesses (such as infectious diseases) requiring compulsory isolation treatment;
* Has received a live vaccine within 30 days prior to the first dose of trial treatment; · · According to the investigator, there may be increased risk associated with participation in the study, or other severe, acute or chronic medical or psychiatric disorders that may interfere with the interpretation of the findings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Approximately 2 months
  Objective response rate by immune related response criteria (irRC), and RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival | up to 24 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | up to 24 months
The disease control rate | up to 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Guozhu,Xie, Guangzhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong